CLINICAL TRIAL: NCT05537480
Title: Correlation of CGM Metrics With OGTT and Pregnancy Outcomes in Pregnant Women With or Without a High Risk for GDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Director, Head of Clinical Trails Department, Principal Investigator, Clinical Professor, Tel-Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 0620-20TLV
Record Dates: First submitted 2021-10-07; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy Complications; Diabetes Mellitus; Hyperglycemic Disorder
MeSH Terms: conditions — Pregnancy Complications; Diabetes Mellitus; Hyperglycemia | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All are blinded to the CGM results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Normal GCT (Other): Women with GCT <140mg/dl
  Interventions: Device: Continuous glucose monitoring device
- Abnormal GCT (Other): Women with GCT >=140mg/dl
  Interventions: Device: Continuous glucose monitoring device

INTERVENTIONS:
Device: Continuous glucose monitoring device — Continuous glucose monitoring device will be worn by participants during several periods.
  Other Names: CGM, DEXCOM PRO G6

SUMMARY:
the aim of the study is to obtain CGM data concomitant with OGTT and to determine what CGM metrics obtained in pregnant women with and without a high risk of GDM correlate best with the diagnostic OGTT (obtained via the 2-step and 1-step approaches).

DETAILED DESCRIPTION:
Study Objectives

Primary Objective:

1. Obtain CGM data concomitant with OGTT to determine what CGM metrics obtained in pregnant women with and without a high risk of GDM correlate best with the diagnostic OGTT (obtained via the 2-step and 1-step approaches)

   Secondary Objectives:
2. Compare GDM diagnosis using the 1-step and 2-step OGTT
3. Obtain CGM data concomitant with OGTT while comparing reproducibility of the 1-step and 2-step methods
4. Determine what CGM metrics obtained concomitant with OGTT correlate best with maternal and fetal outcomes in pregnant women with and without diagnosed GDM
5. Determine how dysglycemia evolves over the third trimester in women with or without diagnosed GDM
6. Compare hyperglycemia determined with CGM to hyperglycemia determined by SMBG in participants diagnosed with GDM
7. Determine what CGM metrics obtained during the third trimester correlate best with maternal and fetal outcomes in pregnant women with and without diagnosed GDM
8. Determine what CGM metrics obtained in pregnant women correlate best with the need for pharmacologic management of GDM Study Devices Dexcom G6 Pro CGM systems blinded to participants. Sample Size Observational. Not powered. The total sample size is up to 280 participants.

the invastigators anticipate enrollment of 280 participants with up to 50 low risk participants and 230 high risk participants. Risk assessment is based on the glucose challenge test results. This should result in 50-80 participants with GDM out of the 230 high risk participants, and allow for 25% dropout for observation throughout the third trimester in the subset of participants Patient Population Pregnant women undergoing screening for GDM Inclusion Criteria To enroll subjects across the glycemic spectrum.

* Pregnant women at high risk for GDM based on GCT results
* Pregnant women at low risk for GDM based on GCT results.
* Had an ultrasound earlier before 12 weeks to confirm gestational age
* Singleton pregnancy Exclusion Criteria • Pregestational diabetes or overt diabetes diagnosed during enrollment
* Concomitant disease or condition that may compromise patient safety or the ability to complete study tasks including and not limited to, severe mental illness, a diagnosed or suspected eating disorder or any uncontrolled long-term medical condition at the investigator's discretion
* Known (or suspected) allergy to medical grade adhesives
* Use of hydroxyurea (a known interferent of CGM) Study Overview Enrollment will occur at 24-28 weeks of gestation after the GCT. After enrollment, two blinded G6 Pro CGM systems will be placed for a 10-day wear period at the arm. Up to 50 women that passed the GCT (glucose <140 mg/dl) will be enrolled. The other approximately 230 women to be enrolled will have hyperglycemia (≥140 mg/dl) on the GCT. All participants will return 2-7days later for either an OGTT and complete corresponding blood draws (including CBC and HbA1C) and fingerstick samples with self-monitoring blood glucose (SMBG) meter at the fasting and 2-hr timepoints of each OGTT. In order to maintain standartization , Subjects will use freestyle lite glucometerto measure SMBG. be randomized at a 1:1 ratio to begin with either the 75-g OGTT or the 100-g OGTT. The data from the initial OGTT will be blinded to the participants unless significant hyperglycemia is detected (75 g HAPO defined: >105 FPG, >200 2hr-PG and 100g defined: >105 FPG, >240 1hr-PG, >200 2hr-PG, >180 3hr-PG). A second OGTT using the alternate glucose content will be performed 3-6 days later and the data will be blinded to participants and the clinicians. This will allow comparison of the diagnostic tests. A subset of 40 participants will be randomized during the initial randomization (10 from the low risk group and 30 from high risk group) will receive the same glucose content in the second OGTT to determine reproducibility of the OGTT. In other words, 20 participants with an initial 75-g OGTT will receive the 75-g dose again at the second OGTT, and 20 participants with an initial 100-g OGTT will receive the 100-g dose again at their second OGTT.

Following the second OGTT the results of the 100-g OGTT will be unblinded (if it was the initial OGTT performed and will be used for diagnostic and management purposes). For those participants that had repeated 75-g OGTT, the results of the initial blinded OGTT will be used for diagnostic and management purposes (after the second OGTT is performed).

Due to the second OGTT, there will be a ~3-day delay in the diagnosys of GDM. This delay has minimal/non-significat ifluence on pregnancy outcome.

The CGM data will be blinded to the patient and clinician and will only be used for research purposes.

Following the OGTT, all 280 participants will have a new CGM placed and participants will be instructed on inserting a CGM system. They will wear a blinded CGM system for 10 days, approximately every other 10-day period through the third trimester until delivery. After each wear session, devices will be sent back to the clinical staff. Medications used to manage GDM and maternal and neonatal outcome data will be collected.

Study Visits Visit 1/Screening & Enrollment (day 0): Participants will complete the informed consent process and complete screening to ensure participant meets inclusion and exclusion criteria. Screening includes GCT with risk assessment based on threshold of 140 mg/dl. Randomization to the different OGTT groups and to the reprodusibility OGTT will be performed. Two CGM systems will be inserted with display blinded.

Patients will be asked to fill a 24-48 hours diet log prior to the first OGTT, thogh it will no be mandatory for the study.

Visit 2/OGTT 1 (day 2 to 7): Study staff will confirm the CGM systems are collecting data. If not, replacement systems will be inserted. Participants will complete either the 75-g or 100-g OGTT and the corresponding blood draws (including CBC and HbA1C). In addition (if possible), fingerstick samples should be obtained with self-monitoed blood glucose (SMBG) at the fasting and 2-hr timepoints of each OGTT. Results will not be provided to the participant but will be reviewed by study staff to confirm there is no overt hyperglycemia requiring unblinding and management of GDM or overt diabetes.

Visit 3/OGTT 2 (day 4 to 10): Study staff will confirm both CGM systems are collecting data. For the subgroup of participants enrolled in the OGTT comparison study (n≤240), participants will complete an OGTT that is the alternate glucose dose provided at Visit 2/OGTT 1, and complete corresponding blood draws and fingersticks per protocol. For the subgroup of participants enrolled in the reproducibility study (n≤40), participants will complete an OGTT that is the same glucose dose provided at Visit 2/OGTT 1.

Visits 2 and 3 will be performed within 2 weeks, and at least 48 hours between them. The third visit will be attempted to be completed prior to 28+6 weeks.

Visit 4/ unblinding OGTT (Day 10): Data from the 100-g OGTT will be unblinded and used for diagnosis by Carpenter & Coustan criteria and management. For participants that had both OGTT using 75-g glucose loads, the initial OGTT will be used for GDM diagnostic purposes using the IADPSG criteria.

In case a participant will complete only one OGTT, due to either technical issues or to personal choice/refussal after completing the first OGTT, she will still remain in the studty. The test that was performed will be unblined and will be used for diagnosis as mentioned above.

Following the OGTT, the CGM sensors will be removed and a new CGM sensor will be deployed by all the participants (whether or not they have GDM) and an additional 3-4 sensors and transmitters will be provided for deployment at home at approximately 3 week intervals. This will allow multiple 10 day wear periods to collect blinded glucose data followed by a 10/11 day breaks off of CGM during the third trimester (objectives 5,7, and 8). The breaks from wearing CGM may help study retention. The CGM data will be blinded to participants and their management will otherwise be usual care for patients with or without GDM. After each wear session, participants will mail back the CGM transmitters to the study staff to download the CGM data. The transmitter should be returned withing 10 days after it is removed.

Optional phone visits: (approximately every 3 weeks): For all participants enrolled through the third trimester, the clinical research team may remind the participant to insert a new CGM and may remotely help participants with deployment issues or other CGM issues. After the wear session, participants may mail back CGM system to study staff so that transmitter is received within 2 weeks for removal.

Data collected • Complete CGM information, (including insertion time/place), GCT, OGTT,(including time/place of measurements taken and brand of blood-glucose meter) HbA1c results.

* Maternal information including: age, height, pre-pregnancy weight, gestational weight gain, mode of conception, number of pregnancies, number of prior deliveries, ethnicity, chronic diseases, smoking habits.
* Pregnancy and delivery information: diagnosis of GDM (including use of insulin or oral agents), length of pregnancy, mode of delivery (and indication for intervention), pregnancy complication, delivery compication (3rd/4th lacerations), shoulder dystocia, LGA, PPH, blood products transfusion.
* Fetal outcome indluding: Gender, weight, apgar score, neonatal hypoglycemia , time in NICU, umbilical cord pH.

Analyses • Correlate basic CGM metrics at week 24-28 with GDM diagnosis by the 75 and 100-g OGTT approaches

* Descriptive statistics of CGM metrics obtained at the time of the OGTT in participants diagnosed with GDM compared to those without GDM
* Compare CGM metrics in participants that need pharmacotherapy to those that don't
* Compare diagnosis by each of the OGTT approaches
* Correlate CGM metrics obtained at the time of the OGTT with maternal and fetal outcomes in women with and without diagnosed GDM (ex: Sung J, et al. AM J Perinatol 2015; 32:461-468)
* Correlate CGM metrics obtained during the third trimester with maternal and fetal outcomes in women with and without diagnosed GDM
* Correlate CGM metrics obtained at the time of the OGTT with CGM metrics obtained during the third trimester
* Compare reproducibility of the diagnostic for the 75 and 100-g OGTT
* Compare dysglycemia determined by CGM compares with dysglycemia determined by SMBG in women diagnosed with GDM
* Compare diagnostic performance (sensitivity, specificity, PPV, NPV) of 1-step vs. 2-step and diagnostic CGM vs. 2-step.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at high risk for GDM based on GCT results
* Pregnant women at low risk for GDM based on GCT results.
* Had an ultrasound earlier before 12 weeks to confirm gestational age
* Singleton pregnancy

Exclusion Criteria:

* Pregestational diabetes or overt diabetes diagnosed during enrollment
* Concomitant disease or condition that may compromise patient safety or the ability to complete study tasks including and not limited to, severe mental illness, a diagnosed or suspected eating disorder or any uncontrolled long-term medical condition at the investigator's discretion
* Known (or suspected) allergy to medical grade adhesives
* Use of hydroxyurea (a known interferent of CGM)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only pregnant women
Enrollment: 280 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Obtain CGM data concomitant with OGTT to determine what CGM metrics obtained in pregnant women with and without a high risk of GDM correlate best with the diagnostic OGTT (obtained via the 2-step and 1-step approaches) | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose

SECONDARY OUTCOMES:
Compare GDM diagnosis using the 1-step and 2-step OGTT | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose
Obtain CGM data concomitant with OGTT while comparing reproducibility of the 1-step and 2-step methods | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose
Determine what CGM metrics obtained concomitant with OGTT correlate best with maternal and fetal outcomes in pregnant women with and without diagnosed GDM | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose
Determine how dysglycemia evolves over the third trimester in women with or without diagnosed GDM | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose
Compare hyperglycemia determined with CGM to hyperglycemia determined by SMBG in participants diagnosed with GDM | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose
Determine what CGM metrics obtained during the third trimester correlate best with maternal and fetal outcomes in pregnant women with and without diagnosed GDM | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose
Determine what CGM metrics obtained in pregnant women correlate best with the need for pharmacologic management of GDM | 2 years
  blood level will be measured of CGM versus self monitoring blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: Liran Hirsh, prof, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Souraski MC, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No